CLINICAL TRIAL: NCT02636231
Title: A Phase II Randomized Controlled Study to Compare Endostar and IMRT vs. IMRT Alone for Locally Recurrent Nasopharyngeal Carcinoma Patients
Brief Title: Endostar for Locally Recurrent Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: JiangXi Province Tumor Hospital (Unknown); The First Affiliated Hospital of Clinical Medicine of G.D.P.U. (Unknown); Second Affiliated Hospital of Nanchang University (Other); First People's Hospital of Foshan (Other); Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); The Affiliated Ganzhou Hospital of Nanchang University (Other); First Affiliated Hospital of Gannan Medical University (Other)
Responsible Party: Principal Investigator, Fei Han, Associate Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NPC201501
Record Dates: First submitted 2015-02-27; First posted 2015-12-21 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Endostar; IMRT; recurrent; NPC
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Recurrence | interventions — Endostatins; endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IMRT and concurrent Endostar (Active Comparator): IMRT and concurrent Endostar (Endostatins) to treat locally recurrent NPC patients; Endostar is to give from the first day of IMRT, 201mg, civ d1-14, q3w for two cycles.
  IMRT is to give GTV 60Gy in 27 fractions.
  Interventions: Drug: Endostatins; Radiation: IMRT
- IMRT alone (Experimental): IMRT alone to treat locally recurrent NPC patients. IMRT is to give GTV 60Gy in 27 fractions.
  Interventions: Radiation: IMRT

INTERVENTIONS:
Drug: Endostatins — Endostar (Endostatins) is to give from the first day of IMRT, 201mg, civ d1-14, q3w for two cycles.
  Other Names: Endostar
  Arms: IMRT and concurrent Endostar
Radiation: IMRT — IMRT is to give GTV 60Gy in 27 fractions.

SUMMARY:
The purpose of this study is to determine whether endostar and IMRT is effective in the treatment of locally recurrent nasopharyngeal carcinoma patients compared with IMRT alone.

DETAILED DESCRIPTION:
Locally recurrent nasopharyngeal carcinoma (NPC) may be salvaged by intensity modulated-radiotherapy (IMRT), but severe late toxicities become the most common reason of death in IMRT salvaged NPC patients.

The aim of this phase II randomized controlled study is to address the efficacy of concurrent Endostar (Endostatins) with IMRT to reduce the occurrence of severe late toxicities compared with IMRT alone for locally recurrent NPC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically or clinically confirmed locally recurrent nasopharyngeal carcinoma;
2. No evidence of distant metastasis
3. More than 1 year from the end of the first course of radiotherapy
4. Male, or female not in the phase of lactating or pregnancy
5. ECOG 0-2
6. Aged 18-70 years old
7. WBC count ≥4×109/L, neutrophile granulocyte count≥1.5×109/L, PLT count ≥100×109/L, Hb ≥9g/L
8. Total bilirubin, AST, ALT≤2.0 times of upper normal limits; creatinine ≤1.5 times of upper normal limits
9. Written informed consort signed

Exclusion Criteria:

1. Only regionally recurrence
2. Evidence of distant metastasis
3. Prior invasive malignancy; noninvasive cancers (For example, carcinoma in situ of the bladder, oral cavity, or cervix are all permissible) are permitted
4. Severe, active co-morbidity
5. Prior anti-tumor treatment after diagnosis of local recurrence
6. MRI was not performed 3 months after the first course of radiotherapy
7. Abnormal function of heart, brain and lungs, etc
8. Lactation or pregnancy
9. Severe nasopharyngeal mucosal necrosis at the diagnosis of local recurrence

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with grade 4-5 late adverse events as assessed by RTOG/EORTC Late Radiation Morbidity Scoring Schema | From 3 months after the end of IMRT to 1 year after the end of IMRT

SECONDARY OUTCOMES:
Number of participants with severe acute toxicities as assessed by CTCAE v3.0 | From the beginning of IMRT to 3 months after the end of IMRT
Overall survival | From the beginning the IMRT to 3 year after the end of IMRT

CONTACTS AND LOCATIONS:
Overall Officials: Fei Han, M.D., Ph.D., Principal Investigator — China: Ethics Committee
Locations (8):
- China (8):
  - First People's Hospital of Foshan, Foshan, Guangdong
  - Cancer Center of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Clinical Medicine of G.D.P.U., Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The Affiliated GanZhou Hospital of NanChang University, Ganzhou, Jiangxi
  - The First Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - JiangXi Province Tumor Hospital, Nanchang, Jiangxi

REFERENCES:
- [Result] Han F, Zhao C, Huang SM, Lu LX, Huang Y, Deng XW, Mai WY, Teh BS, Butler EB, Lu TX. Long-term outcomes and prognostic factors of re-irradiation for locally recurrent nasopharyngeal carcinoma using intensity-modulated radiotherapy. Clin Oncol (R Coll Radiol). 2012 Oct;24(8):569-76. doi: 10.1016/j.clon.2011.11.010. Epub 2011 Dec 29. PMID 22209574
- [Result] Zhang K, Yang S, Zhu Y, Mo A, Zhang D, Liu L. Protection against acute radiation-induced lung injury: a novel role for the anti-angiogenic agent Endostar. Mol Med Rep. 2012 Aug;6(2):309-15. doi: 10.3892/mmr.2012.903. Epub 2012 May 4. PMID 22562140
- [Result] Peng F, Xu Z, Wang J, Chen Y, Li Q, Zuo Y, Chen J, Hu X, Zhou Q, Wang Y, Ma H, Bao Y, Chen M. Recombinant human endostatin normalizes tumor vasculature and enhances radiation response in xenografted human nasopharyngeal carcinoma models. PLoS One. 2012;7(4):e34646. doi: 10.1371/journal.pone.0034646. Epub 2012 Apr 9. PMID 22496834
- [Result] Tong RT, Boucher Y, Kozin SV, Winkler F, Hicklin DJ, Jain RK. Vascular normalization by vascular endothelial growth factor receptor 2 blockade induces a pressure gradient across the vasculature and improves drug penetration in tumors. Cancer Res. 2004 Jun 1;64(11):3731-6. doi: 10.1158/0008-5472.CAN-04-0074. PMID 15172975
- [Result] Tian YM, Guan Y, Xiao WW, Zeng L, Liu S, Lu TX, Zhao C, Han F. Long-term survival and late complications in intensity-modulated radiotherapy of locally recurrent T1 to T2 nasopharyngeal carcinoma. Head Neck. 2016 Feb;38(2):225-31. doi: 10.1002/hed.23880. Epub 2015 May 27. PMID 25244494